CLINICAL TRIAL: NCT03652623
Title: Transgender Youth and PrEP: PK, Safety, Uptake & Adherence
Brief Title: Transgender Youth and PrEP: PK, Safety, Uptake & Adherence - PK Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hektoen Institute for Medical Research (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01MH114753-1; R01MH114753 (NIH)
Record Dates: First submitted 2018-06-25; First posted 2018-08-29 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: HIV/AIDS; Gender; Behavior and Behavior Mechanisms
Keywords: Transgender; Pre-exposure Prophylaxis (PrEP); HIV Prevention; Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC); Cross-sex Hormone Therapy; Adherence; Behavior Change; Gender Affirmation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Coitus; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TDF/FTC and cs-HT (Experimental): Transgender youth will simultaneously take TDF/FTC and cs-HT. TW will take oral estradiol +/- spironolactone and TM will take subcutaneous testosterone. In order to ensure adherence to TDF/FTC, daily DOT procedures will be employed.
  Interventions: Drug: TDF/FTC

INTERVENTIONS:
Drug: TDF/FTC — In Phase 1, a PK study will be conducted to evaluate the differential PK of TDF/FTC in a cohort of transgender youth on cs-HT by conducting a PK trial of daily TDF/FTC among transgender women taking estradiol and transgender men taking testosterone (ages 15-24 years) using video-based directly observed therapy (DOT) to insure daily TDF/FTC adherence and maximize drug exposure.

SUMMARY:
To address the critical scientific gaps in PrEP safety for transgender youth and to plan for appropriate implementation of PrEP in transgender youth communities, the study will be conducted in 3 integrated phases. In Phase 1, a pharmacokinetic (PK) study exploring the interactions of cs-HT for both TW and TM youth on TDF/FTC will be conducted. Simultaneously, in Phase 2, ethnographic data via focus groups (FGs) and in-depth interviews (IDIs) to inform the development of a tailored intervention to improve uptake and adherence to PrEP for transgender youth will be collected. In Phase 3, a small demonstration trial of PrEP use in transgender youth, utilizing the ethnographically developed intervention to improve uptake and adherence, while also monitoring renal and bone safety outcomes will be implemented.

The project has the following important specific aims:

Aim 1: To evaluate the differential PK of TDF/FTC in a cohort of transgender youth on cs-HT by conducting a PK trial of daily TDF/FTC among 24 TW taking estradiol and 24 TM taking testosterone (ages 15-24 years) using video-based directly observed therapy (DOT) to insure daily adherence and maximize drug exposure.

Aim 2: To develop a culturally, developmentally, and gender-affirmative intervention to increase uptake of and adherence to PrEP among TW and TM youth that is grounded in theory (Information-Motivation-Behavioral Skills Model of Behavior Change, Gender Affirmation, Empowerment Theory) and incorporates the PK data from Aim 1. The investigators will conduct FGs with young TW (N=20-30) and TM (N=20-30) and conduct IDIs with participants from the PK study (Total N=10-14). Investigators will solicit continuous input and feedback from TW and TM on the project's Youth Advisory Board.

Aim 3: To conduct a small randomized controlled trial within a PrEP demonstration project comparing the newly developed intervention with standard of care (SOC) in TW (N=50) and TM (N=50) ages 15-24 years.

DETAILED DESCRIPTION:
Transgender women (TW) are one of the most vulnerable populations for acquiring HIV infection, and the scant available data on transgender men (TM) suggests they are also at risk. TW have accounted for only 0.2% of all participants in bio-behavioral HIV prevention trials using pre-exposure prophylaxis (PrEP), and TM have typically not been included. TW and TM adolescents have received even less attention in PrEP trials.

Although tenofovir disoproxil fumarate/emtricitabine (TDF/FTC), the FDA-approved PrEP drug, would not be expected to interact with cross-sex hormone therapy (cs-HT; estradiol and testosterone) based on known mechanisms and data from studies with hormonal contraceptives, there are no data that prove this. Given this lack of data, TW and TM youth on cs-HT have decreased PrEP uptake and adherence due to concerns that PrEP may reduce the effectiveness of cs-HT. To address these critical scientific gaps in PrEP safety for transgender youth and to plan for appropriate implementation, the investigators propose the following study in 3 integrated phases. In Phase 1, the investigators will conduct a PK study exploring the interactions of cs-HT for both TW and TM on TDF/FTC. Simultaneously, in Phase 2, the investigators will collect ethnographic data via focus groups and in-depth interviews to inform the development of a tailored gender-affirmative intervention to improve uptake and adherence to PrEP in transgender youth. In Phase 3, the investigators will conduct a small demonstration trial of PrEP use in TW and TM youth, utilizing the ethnographically developed intervention to improve uptake and adherence, while also monitoring renal and bone safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as a transgender individual [As determined by the two-step process of gender identification whereby potential participants will be asked their gender identity and sex assigned at birth]
* HIV-uninfected by EIA and viral load within 7 days of study entry
* Creatinine clearance ≥ 60 mL/min by Cockroft Gault for ages ≥18 years (Schwartz equation for those <18)
* Willing to comply with all study procedures
* On a stable dose of cs-HT for at least 2 months verified by clinical chart review and willing to not change doses for duration of PK study

Exclusion Criteria:

* Hospitalization within 30 days of study entry (elective procedures okay with team approval)
* Condition (medical, psychological, or social) that, in the opinion of the study investigators, would preclude the participant from completing study-required procedures
* Previous participation in an HIV vaccine study, unless the participant can document placebo arm assignment
* Use of TDF/FTC in the past 3 months

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Self-identification as a transgender individual
Enrollment: 49 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Tenofovir Levels | Baseline and Weeks 0, 1, 2, 3 & 4
  Tenofovir levels in a cohort of transgender youth on cs-HT
Change in Estradiol Levels | Baseline and Weeks 0, 1, 2, 3 & 4
  Estradiol levels in a cohort of transgender youth on cs-HT
Change in Testosterone Levels | Baseline and Weeks 0, 1, 2, 3 & 4
  Testosterone levels in a cohort of transgender youth on cs-HT

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Hosek, PhD, Principal Investigator — Cook County Health
Locations (1):
- University of Colorado, Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yager J, Brooks KM, Brothers J, Mulligan K, Landovitz R, Reirden D, Glenny C, Malhotra M, Anderson PL, Hosek S. Pharmacokinetics of Emtricitabine/Tenofovir Disoproxil Fumarate Among Transgender Adolescents and Young Adults Without HIV Receiving Gender Affirming Hormones. AIDS Res Hum Retroviruses. 2022 Nov;38(11):840-846. doi: 10.1089/AID.2022.0043. Epub 2022 Sep 7. PMID 35943868
- [Derived] Yager J, Brooks KM, Brothers J, Mulligan K, Landovitz RJ, Reirden D, Malhotra M, Glenny C, Harding P, Powell T, Anderson PL, Hosek S. Gender-Affirming Hormone Pharmacokinetics Among Adolescent and Young Adult Transgender Persons Receiving Daily Emtricitabine/Tenofovir Disoproxil Fumarate. AIDS Res Hum Retroviruses. 2022 Dec;38(12):939-943. doi: 10.1089/AID.2022.0044. Epub 2022 Aug 9. PMID 35815468